CLINICAL TRIAL: NCT00003819
Title: Vaccination of Prostate Cancer Patients With Thompson-Friedenreich [TF(c)]-KLH Conjugate Plus the Immunological Adjuvant QS21: A Trial Comparing TF(c)-KLH Doses
Brief Title: Vaccine Therapy Plus QS21 in Treating Patients With Progressive Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-048; P30CA008748 (NIH); MSKCC-98048; NCI-G99-1510
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — saponin QA-21V1; Thomsen-Friedenreich antigen; keyhole-limpet hemocyanin

ARMS (1):
- vaccine (Experimental): This is a dose escalation study. Patients receive TF(c)-KLH conjugate with adjuvant QS21 subcutaneously weekly for 3 weeks, then once during weeks 7 and 19. Cohorts of 5 patients each receive escalating doses of TF(c)-KLH vaccine until the optimal dose, based on antibody response, is reached. Patients are followed monthly for 6 months, then every 3 months for 1 year.
  Interventions: Biological: QS21; Biological: TF(c)-KLH conjugate vaccine; Biological: Thomsen-Friedenreich antigen; Biological: keyhole limpet hemocyanin

INTERVENTIONS:
Biological: QS21
Biological: TF(c)-KLH conjugate vaccine
Biological: Thomsen-Friedenreich antigen
Biological: keyhole limpet hemocyanin

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy given with QS21 in treating patients who have progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the optimal dose of Thompson-Friedenreich [TF(c)]-keyhole limpet hemocyanin (KLH) conjugate plus adjuvant QS21 that induces an antibody response in patients with prostate cancer. II. Determine the safety of the TF(c)-KLH conjugate prepared using an MBS heterobifunctional linker plus QS21. III. Assess postimmunization changes in prostate specific antigen levels and other objective parameters of disease in these patients.

OUTLINE: This is a dose escalation study. Patients receive TF(c)-KLH conjugate with adjuvant QS21 subcutaneously weekly for 3 weeks, then once during weeks 7 and 19. Cohorts of 5 patients each receive escalating doses of TF(c)-KLH vaccine until the optimal dose, based on antibody response, is reached. Patients are followed monthly for 6 months, then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven progressive prostate cancer after primary therapy Radiographic changes OR PSA at least 1.0 ng/mL and rising after prostatectomy OR PSA at least 2.0 ng/mL and rising after radiotherapy OR PSA rising 50% during intermittent hormonal therapy No metastatic disease by radiography No active CNS or epidural tumor Registered on MSKCC-9040

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 6 months Hematopoietic: WBC at least 3500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL OR SGOT less than 3.0 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No New York Heart Association class III/IV cardiac disease Pulmonary: No severe debilitating pulmonary disease Other: No other active malignancy within 5 years except nonmelanomatous skin cancer No infection requiring antibiotics No narcotic dependent pain No positive stool guaiac excluding hemorrhoids No radiation induced proctitis No allergy to seafood

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 2 weeks since change in hormonal therapy (except to maintain castrate levels of testosterone), including prednisone or dexamethasone At least 8 weeks since prior suramin and/or serum concentration of suramin must be less than 50 micrograms/mL (replacement hydrocortisone allowed) Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No concurrent therapy to only measurable lesion Surgery: See Disease Characteristics No concurrent surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1998-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
response | 2 years

SECONDARY OUTCOMES:
safety | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States